CLINICAL TRIAL: NCT05924685
Title: Prospective Randomized Trial of Everolimus Replacing MMF/MP Acid by the RECOVAC Consortium to Increase VACcine Response in Kidney Transplant Patients
Brief Title: PREPARE-iVAC Trial
Acronym: PREPARE-iVAC
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Medical Center Groningen (Other)
Collaborators: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other); Radboud University Medical Center (Other); Erasmus Medical Center (Other); UMC Utrecht (Other); Leiden University Medical Center (Other); Maastricht University Medical Center (Other); ZonMw: The Netherlands Organisation for Health Research and Development (Other); Dutch Kidney Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 11442; 2023-503894-39-00 (Other: EUCTnumber)
Record Dates: First submitted 2023-06-20; First posted 2023-06-29 (Actual); Last update posted 2024-03-04 (Actual); Status verified 2024-03

CONDITIONS: COVID-19 Vaccines; Varicella Zoster Vaccine; Vaccine Response; Immunosuppression
Keywords: Kidney Transplant Recipients; COVID-19 vaccines; Everolimus; Mycophenolate Mofetil; Varicella Zoster Vaccine
MeSH Terms: interventions — heterologous prime boost COVID-19 vaccination

STUDY DESIGN:
Intervention Model Description: Participants will be 1:1 randomised to:
  1. Continue immunosuppressive therapy with MMF/MPA
  2. Replace immunosuppressive therapy with MMF/MPA by everolimus
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Continue immunosuppressive therapy with MMF/MPA (Active Comparator): Kidney transplant recipients with maintenance therapy, receiving the monovalent Omicron XBB.1.5 COVID-19 mRNA vaccine (Comirnaty, I.M.). Optional to receive the Recombinant Zoster Vaccine (Shingrix, I.M.).
  Interventions: Biological: COVID-19 vaccination
- Replace immunosuppressive therapy with MMF/MPA by everolimus (Active Comparator): Kidney transplant recipients replacing MMF/MPA by everolimus for at least six weeks, receiving the monovalent Omicron XBB.1.5 COVID-19 mRNA vaccine (Comirnaty, I.M.). Optional to receive the Recombinant Zoster Vaccine (Shingrix, I.M.).
  Interventions: Biological: COVID-19 vaccination

INTERVENTIONS:
Biological: COVID-19 vaccination — Vaccination
  Other Names: the monovalent Omicron XBB.1.5 COVID-19 mRNA vaccination

SUMMARY:
Objective: To investigate whether replacement of MMF/MPA by everolimus in kidney transplant recipients results in superior immunogenicity of COVID-19 vaccination as measured by neutralizing antibody titer against the Omicron XBB.1.5 strain.

Trial design: Multicentre, open-label randomized controlled clinical trial, for a duration of at least 10 weeks with an optional extension to 18 weeks.

Trial population: Kidney transplant recipients, 18 years or older, who are at least 6 months after transplantation, with a functioning kidney transplant, using MMF/MPA in combination with at least one other immunosuppressant including a calcineurin inhibitor (CNI), with at least 3 previous COVID-19 vaccinations (=basic COVID-19 immunisation).

Interventions:

Patients will be randomized into one of two equally sized groups, with either continuation of their current immunosuppressive regimen including MMF/MPA or replacement of MMF/MPA by everolimus during at least six weeks before until four weeks after the last vaccination. Patients will receive a repeated COVID-19 vaccination with the monovalent Omicron XBB.1.5 vaccine, 28 days thereafter they can opt to also receive two herpes zoster vaccinations with the Recombinant Zoster Vaccine (RZV) with an interval between the first and second dose of 28 days.

Main trial endpoints:

The neutralizing antibody titer against the Omicron XBB.1.5. strain 28 days after monovalent Omicron XBB.1.5 COVID-19 vaccination in patients continuing MMF/MPA compared to patients who switched to everolimus.

Secondary trial endpoints:

* SARS-CoV-2 specific anti-S1 antibody level at 28 and 56 days after COVID-19 vaccination
* Varicella zoster specific anti-gE antibody level 28 days after 1st and 2nd herpes zoster vaccination
* SARS-CoV-2 specific T-cell response 28 days after COVID-19 vaccination
* Varicella zoster specific T-cell response 28 days after 2nd herpes zoster vaccination
* Safety in terms of incidence of acute rejection, kidney function decline, SAEs, AESIs and solicited local and systemic AEs after COVID-19 and herpes zoster vaccination

DETAILED DESCRIPTION:
Rationale: The immunogenicity after vaccination against SARS-CoV-2 and other pathogens is diminished in kidney transplant recipients. This patient group therefore remains extremely vulnerable for viral infections despite vaccination. This impaired immune response is related to the use of immunosuppressive agents, especially Mycophenolate Mofetil/Mycophenolic Acid (MMF/MPA). Patients that use everolimus instead of MMF/MPA elicit a higher immune response after vaccination.

Objective

Primary objective:

To investigate whether replacement of MMF/MPA by everolimus in kidney transplant recipients results in superior immunogenicity of COVID-19 vaccination as measured by neutralizing antibody titer against the Omicron XBB.1.5 strain.

Secondary objectives:

* To investigate whether replacement of MMF/MPA by everolimus in kidney transplant recipients results in superior humoral immunogenicity of

  * COVID-19 vaccination as measured by SARS-CoV-2 specific anti-S1 antibody levels
  * herpes zoster vaccination as measured by varicella zoster specific anti-gE antibody levels
* To investigate whether replacement of MMF/MPA by everolimus in kidney transplant recipients results in superior cellular immunogenicity of

  * COVID-19 vaccination as measured by SARS-CoV-2 specific T-cell response
  * herpes zoster vaccination as measured by varicella zoster specific T-cell response
* To evaluate safety of replacement of MMF/MPA by everolimus in terms of

  * incidence of treated acute rejection, kidney function decline, incidence of serious adverse events (SAEs)
  * incidence of adverse events of special interest (AESI) of immunosuppression
  * incidence of solicited adverse events (AEs) of COVID-19 vaccination
  * incidence of solicited AEs of herpes zoster vaccination

This is a multicentre, open-label, controlled, randomized study to evaluate replacement of MMF/MPA by everolimus in KTR on immunogenicity and safety after vaccination.

The seven participating study sites are Amsterdam UMC, Erasmus MC, Leiden UMC, Maastricht UMC+, Radboudumc, UMC Groningen and UMC Utrecht.

At the first study visit, eligibility for study participation will be checked, blood will be drawn, and participants will subsequently be 1:1 randomised to:

1. Continue immunosuppressive therapy with MMF/MPA
2. Replace immunosuppressive therapy with MMF/MPA by everolimus

After randomisation, the study will continue in 2 parts:

Part 1 - Run-in and COVID-19 vaccination (≥6 weeks + 28 days) The aim of this phase is to first ensure complete washout of MMF/MPA and attaining optimal trough levels of everolimus in patients randomized to everolimus.

To monitor tolerability, safety and trough levels, participants will be invited at week 1 and week 3 after randomisation for a blood withdrawal and spot urine collection.

At least 6 weeks after randomisation, patients will receive the COVID-19 vaccination (=baseline visit). After 28 days patients will be invited for a study visit for blood withdrawal.

Part 2 (optional) - Herpes zoster vaccination (+56 days) Patients that opted to participate in this part of the study will continue their randomised treatment for the next 56 days. During this period patients will receive 2 herpes zoster vaccinations with an interval of 28 days between each vaccination. At 28 days after the second vaccination patients will be invited for the last study visit for blood withdrawal.

After completion of the study (either 28 days after COVID-19 vaccination or 28 days after the last herpes zoster vaccination) patients will be offered the option to continue everolimus instead of MMF/MPA as part of shared clinical decision making.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* ≥6 months after kidney transplantation
* Maintenance immunosuppressive therapy consisting of either triple or dual therapy including MMF/MPA with a minimum daily dose of 1000 mg (MMF) or 720 mg (MPA) and a CNI
* Eligible for the vaccinations as described by the instructions of the manufacturers of the vaccines (e.g. received 3 previous COVID-19 vaccinations as part of the primary COVID-19 immunisation)
* Capable of understanding the purpose and risks of the study, fully informed and given written informed consent (signed informed consent form has been obtained)
* Willing to adhere to the protocol and be available during the study period

Exclusion Criteria:

* Previous CNI trough levels not sufficient according to the discretion of the treating physician
* More than two previous kidney transplantations
* Calculated level of panel reactive antibodies prior to last transplantation above 85%
* Evidence of DSAs
* Signs of acute rejection during the preceding year
* Multi-organ transplant recipient
* History of severe adverse reaction associated with a vaccine and/or severe allergic reaction (e.g. anaphylaxis) to any component of the study intervention(s)
* Contra-indications for use of everolimus according to the opinion of the treating physician
* Active COVID-19 disease
* Active malignancy, except non-melanoma skin cancer
* Inherited immune deficiency
* Infection with Human Immunodeficiency Virus (HIV)
* Administration of T-cell, B-cell, or plasma cell depleting antibodies during the last 6 months
* Bleeding diathesis or condition associated with prolonged bleeding that would, in the opinion of the investigator, contraindicate intramuscular injection
* Subjects with severe systemic infections, current or within the two weeks prior to randomisation
* Subjects with severe restrictive or obstructive pulmonary disorders
* Subjects with severe hypercholesterolemia or hypertriglyceridemia that cannot be controlled
* Subjects with white blood cell (WBC) count ≤ 2,000/mm3 or with platelet count ≤ 50,000/mm3 at last outpatient clinic visit
* Proteinuria > 1 gram/day at last outpatient clinic visit
* Simultaneous participation in another interventional study that will likely influence the study outcomes
* Subject who are actively trying to get pregnant or are pregnant

Additional exclusion criteria for Part 2:

* Active varicella or herpes zoster disease
* Herpes zoster vaccination with the live attenuated vaccine (Zostavax) or varicella vaccination (Provarivax) during the conduct of the study
* Previous herpes zoster vaccination with the RZV

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2023-08-22 (Actual); Primary Completion 2023-12-29 (Actual); Study Completion 2024-02-27 (Actual)

PRIMARY OUTCOMES:
Virus-neutralizing capacity of SARS-CoV-2 antibodies | 28 days after COVID-19 vaccination
  The neutralizing antibody titer against the Omicron XBB.1.5 strain

SECONDARY OUTCOMES:
SARS-CoV-2 antibody concentration | 28 days after COVID-19 vaccination
  SARS-CoV-2 specific anti-S1 antibody concentrations in serum
SARS-CoV-2 specific T-cell response | 28 days after COVID-19 vaccination
  SARS-CoV-2 specific T-cell response
Varicella Zoster specific antibodies | 28 days after second Varicella Zoster vaccination
  Concentrations of Varicella Zoster specific anti-gE antibodies
Varicella Zoster specific T-cell Response | 28 days after second Varicella Zoster vaccination
  Varicella Zoster specific T-cell response
Solicited local and systemic adverse events | Within 7 days after vaccination
  Percentage of participants reporting local reactions (pain at the injection site, redness and swelling) and systemic events (fever, fatigue, headache, chills, vomiting, diarrhea, new of worsened muscle pain, and new or worsened joint pain) after COVID-19 and both Varicella Zoster vaccines administration
Serious adverse events | Within 84 days after COVID-19 vaccination
  Percentage of participants with serious adverse events after COVID-19 and both Varicella Zoster vaccines administration, with special interest in treatment of acute rejection.
Safety of kidney transplant | From enrollment to 84 days after COVID-19 vaccination
  Change in estimated glomerular filtration rate and proteinuria during the study including creatinine measurements in blood and protein measurements in spot urine.

OTHER OUTCOMES:
Relationship between previous COVID-19 infection and immune responses | 28 days after vaccination
  The association between immunological outcomes and the timing of a previous COVID-19 infection and COVID-19 severity will be investigated
Virus neutralizing capacity of SARS-CoV-2 antibodies | 28 days after COVID-19 vaccination
  Neutralizing antibody titers against the most common SARS-CoV-2 variant at the moment of study conduct
Delayed SARS-CoV-2 antibody response | 56 days after COVID-19 vaccination
  A potential delayed humoral response after COVID-19 vaccination will be tested by comparing anti-S1 antibody levels at 56 days and 28 days after vaccination
Relationship between baseline clinical features and immune responses | 28 days after vaccination
  Compare/relate baseline clinical features and antibody/T cell responses to the level of induced antibody and T cell responses after vaccination.

CONTACTS AND LOCATIONS:
Overall Officials: Jan-Stephan F Sanders, MD PhD, Principal Investigator — University Medical Center Groningen
Locations (7):
- Netherlands (7):
  - Radboud University Medical Center, Nijmegen, Gelderland
  - Maastricht University Medical Center, Maastricht, Limburg
  - Amsterdam University Medical Center, Amsterdam, North Holland
  - Leiden University Medical Center, Leiden, South Holland
  - Erasmus Medical Center, Rotterdam, South Holland
  - University Medical Center Groningen, Groningen
  - University Medical Center Utrecht, Utrecht

IPD SHARING:
Plan to Share IPD: No
The data of this study will be available from the principal investigator, upon reasonable request.